CLINICAL TRIAL: NCT01035385
Title: Phase III Study to Compared Preoperative and Postoperative With FOFLOX4 Chemotherapy and Postoperative With FOFLOX4 Chemotherapy in Patients With Resectable Liver Metastasis From Colorectal Cancer
Brief Title: Compare FOFLOX4 in Preoperative and Postoperative and Postoperative in Resectable Liver Metastasis Colorectal Cancer (MCC)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Feng Lin/Gastrointestinal Surgery, Guangdong General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VORP019
Record Dates: First submitted 2009-12-16; First posted 2009-12-18 (Estimated); Last update posted 2009-12-18 (Estimated); Status verified 2009-09

CONDITIONS: Colorectal Cancer; Liver Metastasis
Keywords: FOFLOX4; resectable liver metastasis from colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FOFLOX4,resectable liver metastasis from CRC (Experimental)
  Interventions: Drug: FOFLOX4

INTERVENTIONS:
Drug: FOFLOX4 — FOLFOX4:Oxaliplatin 85mg/m2 ivgtt d1 2hr calcium leucovorin:200mg/m2 ivgtt d1 d2 2hr fluorouracil:400mg/m2 iv d1 d2 fluorouracil:600mg/m2 civ d1 d2 22hr 2 weeks repeated one cycles

SUMMARY:
This study is a multicenter, open-label, randomized ,controlled phase III study to compare preoperative and postoperative with FOFLOX4 chemotherapy and postoperative with FOFLOX4 chemotherapy in patients with resectable liver metastasis from colorectal cancer.

DETAILED DESCRIPTION:
To investigate the three-year progression free survival (PFS) advantage of FOLFOX4 in the treatment of resectable metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Resectable liver metastasis from colorectal cancer(the distance from the tumor lower edge to anal more than 12cm),no visible extrahepatic metastatic tumors. Curable by resection, as determined by a surgeon and imaging physicians. The minimum of the liver metastases needs ≥2cm. Patients can be recruited if meet the conditions about:

   * Primary tumor had been removed of the metachronous liver metastasis patients and no residue from the eyes or microscope.
   * Primary tumor has been removed more than 1 month of the simultaneous liver metastasis patients.
2. Age of≥18 and ≤80
3. ECOG≤2
4. Signed written informed consent

Exclusion Criteria:

1. Peripheral neuropathy(CTC>1)
2. Had a neurological or mental disorders
3. Active infection
4. Allergy to Platinum-based and other drugs
5. Other acute diseases including infection, heart-disease(CHF, stable or unstable angina)
6. Pregnant or nursing patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2009-09; Primary Completion 2012-10 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
progression free survival (PFS) | 3 years

SECONDARY OUTCOMES:
response rate, incidence of postoperative complications,pathological response rate,R0 resection rate, 5-year overall survival,duration of disease control | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Feng Lin, Dr, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China